CLINICAL TRIAL: NCT07132749
Title: A Prospective, Observational, Multicenter Cohort Study Evaluating the Efficacy and Safety of NEPA (Netupitant/Palonosetron) in Patients With HER2-positive or HER2-low Advanced Breast Cancer Treated With T-DXd
Brief Title: NEPA in Patients With HER2-positive or HER2-low Advanced Breast Cancer Treated With T-DXd
Acronym: PRO-NEPA
Status: Enrolling by invitation | Type: Observational
Sponsor: Yeon Hee Park (Other)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor-Investigator, Yeon Hee Park, professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: 2025-04-119
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Patients With HER2-positive Advanced Breast Cancer Treated With T-DXd; Patients With HER2-low Advanced Breast Cancer Treated With T-DXd
Keywords: HER2-positive; HER2-low; advanced breast cancer; T-DXd; NEPA; netupitant/palonosetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: advanced breast cancer patients receiving at least 2 cycles of T-DXd.

SUMMARY:
This clinical trial is a prospective, observational, multicenter cohort study evaluating the efficacy and safety of NEPA (netupitant/palonosetron) in patients with HER2-positive or HER2-low advanced breast cancer treated with T-DXd

DETAILED DESCRIPTION:
The observation period of this study is until the discontinuation after administration of T-Dxd or until 8 Cycle.

* Acute phase: 0 -24 hours after T-DXd administration
* Delayed phase: >24-120 hours after T-DXd administration
* Overall phase: 0-120 hours after T-DXd administration
* Long-delayed phase: >120-504 hours
* Extended overall phase: 0-504 hours

Primary objectives: to evaluate the efficacy and safety of NEPA for CINV prevention in advanced breast cancer patients receiving at least 2 cycles of T-DXd across all defined assessment periods (acute, delayed, overall, long-delayed, and extended overall phases).

ELIGIBILITY:
Inclusion Criteria:

1. Age >19 years
2. Histologically confirmed breast cancer with metastatic or locally advanced breast cancer not amenable to definitive surgery, with or without measurable disease
3. Stage IV breast cancer at initial diagnosis (de novo) or progression at distant metastatic sites following curative surgery
4. HER2-positive breast cancer (HER2 IHC 3+ or IHC 2+/ISH-positive) or HER2-low breast cancer (HER2 IHC 2+/ISH-negative or HER2 IHC 1+), as defined by the ASCO/CAP guidelines
5. ECOG performance status 0-2
6. Patients who are scheduled to initiate their first cycle of T-DXd therapy
7. Patients who are scheduled to receive netupitant/palonosetron (NEPA) for the prevention of acute and delayed CINV according to the approved indications and dosage instructions
8. Patients who agree to use highly effective contraception methods or not of childbearing potential. Highly effective contraception methods include:

   A. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

   B. Total hysterectomy (surgical removal of the uterus and cervix) or tubal ligation (getting your "tubes tied") at least six weeks before taking study treatment.

   C. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.

   D. Combination of the following:

   I. Placement of an intrauterine device (IUD) or intrauterine system (IUS) II. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
9. Written informed consent

Exclusion Criteria:

1. Patients who experienced nausea and/or vomiting within 7 days prior to the first cycle of T-DXd treatment
2. Leptomeningeal metastasis and/or brain metastasis
3. Patients with hypersensitivity to any components of the drug or 5-HT3 receptor antagonists.
4. Pregnant women or those suspected of being pregnant, as well as breastfeeding mothers.
5. Any illness or condition that, in the opinion of the Investigator, may pose unwarranted risks in administering T-DXd or NEPA to the patient.
6. Patients requiring treatment with steroids, antiemetics, benzodiazepines, antipsychotics, or other contraindicated drugs, including but not limited to pimozide, terfenadine, astemizole, cisapride, rifampin, carbamazepine, phenytoin, ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, fluvoxamine, SSRIs, SNRIs, ritonavir, or nelfinavir.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had not been previously treated with T-DXd and are scheduled to receive their first cycle of T-DXd with NEPA
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR: no emesis and no rescue medication) | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  CR during the long-delayed phase(>120-504 hours)

SECONDARY OUTCOMES:
Complete response (CR: no emesis and no rescue medication) | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  CR during the acute phase (0-24 hours), delayed phase (>24-120 hours), overall phase (0-120 hours), extended overall phase (0-504 hours)
Complete control (CC: no emesis, no rescue medication and no or mild nausea) | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  CC during the acute phase (0-24 hours), delayed phase (>24-120 hours), overall phase (0-120 hours), long-delayed phase (>120-504 hours), and extended overall phase (0-504 hours)
Total control (TC: no emesis, no rescue medication and no nausea) | At the end of first Cycle 2 of T-DXd (each cycle is 28 day), assessed up to 6 weeks
  TC during the acute phase (0-24 hours), delayed phase (>24-120 hours), overall phase (0-120 hours), long-delayed phase (>120-504 hours), and extended overall phase (0-504 hours)
No significant nausea (NSN: defined as no or mild nausea) | At the end of first Cycle 2 of T-DXd (each cycle is 28 day), assessed up to 6 weeks
  NSN during the acute phase (0-24 hours), delayed phase (>24-120 hours), overall phase (0-120 hours), long-delayed phase (>120-504 hours), and extended overall phase (0-504 hours
No nausea | At the end of first Cycle 2 of T-DXd (each cycle is 28 day), assessed up to 6 weeks
  No nausea during the acute phase (0-24 hours), delayed phase (>24-120 hours), overall phase (0-120 hours), long-delayed phase (>120-504 hours), and extended overall phase (0-504 hours)
CR rate | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  Daily CR rate
NSN rate | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  Daily NSN rate
no nausea rate | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  Daily no nausea rate
Proportion of patients who receive rescue medications | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  Proportion of patients who receive rescue medications
Proportion of patients undergoing T-DXd dose delay | At the end of first documented progression or first Cycle 8 of T-DXd (each cycle is 28 days), assessed up to 24 weeks
  Proportion of patients undergoing T-DXd dose delay due to nausea and/or vomiting
Proportion of patients requiring permanent discontinuation | At the end of first documented progression or first Cycle 8 of T-DXd (each cycle is 28 days), assessed up to 24 weeks
  Proportion of patients requiring permanent discontinuation of T-DXd due to nausea and/or vomiting
Health-related quality of life (EQ-5D-5L) | At the end of first documented progression or first Cycle 8 of T-DXd (each cycle is 28 days), assessed up to 24 weeks
  1. Range of EQ-5D index Minimum-Maximum Range: approx.-0.28 to -0/17 ~ 1,000
  2. Range of EQ VASMinimum-Maximum Range: 0~100 *The higher to score, the better the health status.
FACIT Fatigue | At the end of first documented progression or first Cycle 8 of T-DXd (each cycle is 28 days), assessed up to 24 weeks
  Proportion of patients experiencing fatigue and severity of fatigue (FACIT Fatigue) (1) Range of FACIT Fatigue scale Minimum-Maximum Range 0~52
  *Higher score indicate less fatigue and better health status.
CTCAE v5.0 | At the end of first documented progression or first Cycle 8 of T-DXd (each cycle is 28 days), assessed up to 24 weeks
  Safety evaluated according to CTCAE v5.0, higher scores mean a worse outcome
Daily rescue medication rate | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  Daily rescue medication rate
Duration of rescue medication | At the end of first Cycle 2 of T-DXd (each cycle is 28 days), assessed up to 6 weeks
  Duration of rescue medication

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided later.